CLINICAL TRIAL: NCT03500068
Title: Establishing Organoids From Metastatic Pancreatic Cancer Patients, the OPT-I Study
Acronym: OPT-1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, J.W. Wilmink, M.D. PhD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2017-202
Record Dates: First submitted 2018-04-09; First posted 2018-04-17 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Carcinoma, Pancreatic Ductal
Keywords: Pancreatic cancer; Organoids
MeSH Terms: conditions — Carcinoma, Pancreatic Ductal; Pancreatic Neoplasms | interventions — Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: biopsies & blood analyses — They will take blood and a biopsy from the metastase in the patient

SUMMARY:
Rationale: Pancreatic adenocarcinoma is a malignancy with a poor prognosis. Resection is the only curative option and still 5-year survival rate is less than 10 percent. However, most patients present with advanced disease and are provided with palliative care. The nature of the tumour and the intense stromal reaction around the tumour cells leave pancreatic adenocarcinoma relatively insensitive to chemotherapeutics. Current models, such as cell lines or patient derived xenografts, cannot provide predictive information in a clinically relevant timeframe. Organoids and organotypic culture systems have emerged as promising new culturing techniques that maintain some of the complexity of the tumour. As most patients are ineligible for tumour resection, this project will focus on metastases and will generate organoids from that tissue. Using a combination of organoids and organotypic systems, treatment (non)response can be predicted, which may provide a personalized treatment setting for patients with advanced pancreatic adenocarcinoma.

DETAILED DESCRIPTION:
Rationale: Pancreatic adenocarcinoma is a malignancy with a poor prognosis. Resection is the only curative option and still 5-year survival rate is less than 10 percent. However, most patients present with advanced disease and are provided with palliative care. The nature of the tumour and the intense stromal reaction around the tumour cells leave pancreatic adenocarcinoma relatively insensitive to chemotherapeutics. Current models, such as cell lines or patient derived xenografts, cannot provide predictive information in a clinically relevant timeframe. Organoids and organotypic culture systems have emerged as promising new culturing techniques that maintain some of the complexity of the tumour. As most patients are ineligible for tumour resection, this project will focus on metastases and will generate organoids from that tissue. Using a combination of organoids and organotypic systems, treatment (non)response can be predicted, which may provide a personalized treatment setting for patients with advanced pancreatic adenocarcinoma.

Objective: To develop a model system and infrastructure to individualize the treatment of patients with advanced pancreatic adenocarcinoma. Additionally, we aim to identify predictors of therapy (non)response.

Study design: Observational laboratory studies (with DNA/RNA isolation, RNA sequencing, cell culturing, organoid culturing and xenografting) will be performed with tumour specimens. These organoids will be stored for future research.

Study population: All adult patients (> 18 years) with (a suspicion of) advanced pancreatic adenocarcinoma

Main study parameters/endpoints: The development of organoids from biopsies of metastases or primary tumour tissue of pancreatic cancer that correlate with clinical response. These models are then analysed for the expression of bio markers in organoid, organotypic and xenograft models. DNA/RNA profiles will be correlated to clinical and pathological characteristics such as therapy response, survival and TNM classification.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Participating in this study requires a biopsy from the patient. The material will be obtained from the biopsy required for diagnosis or the patient is asked for consent for an additional tumor biopsy not required for diagnosis. The study could benefit patients as their organoids can be used to assess efficacy of first-line treatment and when necessary may provide an advice for second-line treatment options. Additionally, patients may benefit in the future, if biomarkers are found to predict therapy (non)response.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years
* Diagnosed with locally advanced pancreatic cancer or metastatic pancreatic cancer
* Able to understand the information given
* WHO 0-2

Exclusion Criteria:

* Unfit for biopsies & blood analyses
* Not able to give informed consent (language, intellectual capacities, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-09-04 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Developing organoids from advanced pancreatic cancer patients that predict non response or response | 2 months
  To assess whether there is a correlation between no response in patients and no response in organoids, a goodness of fit will be determined with Pearson's X2 test. Depending on the available data, the second scenario will be analysed similarly.
  When organoids cannot be established from biopsy material, then this will be recorded and linked to clinical parameters.

SECONDARY OUTCOMES:
Functional studies will be done with the patient derived organoids to find biomarkers that correlate with response in organoids and patients. | 2 months
  Similarly to our primary study parameter, the value of prediction for a biomarker will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Academic Medical Center, Medical Oncology, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No